CLINICAL TRIAL: NCT02816580
Title: PTMDP (Post-translational Modification Derived Products) as Markers of Frailty in Elderly Subjects
Brief Title: Biological MArkers of FRAilty in Elderly Subjects
Acronym: MAFRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO14057
Record Dates: First submitted 2016-06-17; First posted 2016-06-28 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2022-02

CONDITIONS: Elderly Persons
MeSH Terms: interventions — Blood Specimen Collection

ARMS (1):
- elderly subjects (Experimental)
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection

SUMMARY:
Epidemiological data from Europe have shown that around 30% of subjects aged over 65 years of age are pre-frail, and 15% are frail. Recent research has demonstrated that identifying frailty and implementing preventive measures can help to slow cognitive decline. Screening and treating frailty seem to be a good start towards preventing dependency.

On the premise that this frailty is the result of more pronounced tissue alterations in certain elderly subjects, assessment of post-translational modification derived products (PTMDP) represents an innovative evaluation method. These include advanced glycation end-products (AGE), and carbamylation-derived products (homocitrulline). Indeed, the intensity of these modifications increases with ageing, and assessing the products resulting from these alterations could show the existence of differences according to frailty status. This would make it possible to adapt treatment accordingly in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

* With social security coverage
* Accept to participate in the study and sign informed consent for the study and for the collection of biological samples

Exclusion Criteria:

- < 65 yo

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 254 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
post-translational modification derived-products (PTMDP) quantification by Multidimensional Chromatography Coupled withTandem Mass Spectrometry (LC/LC-MS/MS) | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Mahmoudi R, Jaisson S, Badr S, Jaidi Y, Bertholon LA, Novella JL, Gillery P. Post-translational modification-derived products are associated with frailty status in elderly subjects. Clin Chem Lab Med. 2019 Jul 26;57(8):1153-1161. doi: 10.1515/cclm-2018-1322. PMID 30817296